CLINICAL TRIAL: NCT06581302
Title: Accelerated 100Hz Magnetic Seizure Therapy for Psychotic Disorders
Brief Title: Magnetic Seizure Therapy for Psychotic Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jijun Wang, Professor of Department of Psychiatry, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-TX-002
Record Dates: First submitted 2024-08-15; First posted 2024-09-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Psychotic Disorders
Keywords: Magnetic Seizure Therapy (MST); psychotic disorders; longitudinal study
MeSH Terms: conditions — Psychotic Disorders | interventions — Risperidone; Aripiprazole; Quetiapine Fumarate; Amisulpride; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic seizure therapy plus antipsychotics (Experimental): The patients will receive antipsychotic drugs plus MST during the first 2 weeks.
  A TwinCoil of MagPro XP will be positioned centrally over the frontal cortex in the midline position. The output power of MagPro XP is set to 100%, and stimulation frequency is 100 Hz. For MST titration, the first step is given at a 5-second train duration; if there is no seizure, the duration is increased to 10 seconds with a maximum limit of 10 seconds. The subsequent MST treatment will be maintained at 10 seconds. This procedure will be carried out under anesthesia.
  A total of up to 10 treatments will be administered to participants, usually five times a week, for 2 weeks.
  Interventions: Device: Magnetic seizure therapy by Magnetic stimulator
- antipsychotic drugs (Active Comparator): The patients will receive second-generation antipsychotic drugs without MST or ECT during the first 2 weeks.
  Interventions: Drug: Antipsychotic medications (such as olanzpine, risperidone, aripiprazole, quetiapine, amisulpride, etc)

INTERVENTIONS:
Device: Magnetic seizure therapy by Magnetic stimulator — The seizure is induced by Magnetic stimulator of MagPro MST(XP)，MagVenture A/S, Farum, Denmark. It is administered in combinations with antipsychotic medications
  Other Names: Seizure therapy
  Arms: Magnetic seizure therapy plus antipsychotics
Drug: Antipsychotic medications (such as olanzpine, risperidone, aripiprazole, quetiapine, amisulpride, etc) — It mainly includes second-generation antipsychotic medications, such as olanzpine, risperidone, aripiprazole, quetiapine, amisulpride, etc, but except clozapine.
  Other Names: antipsychotics
  Arms: antipsychotic drugs

SUMMARY:
This trial aims to evaluate the efficacy and safety of Magnetic Seizure Therapy (MST) as an augmentation of antipsychotic medications for psychosis.

DETAILED DESCRIPTION:
Psychosis is recognized as one of the largest contributors to nonfatal health loss, and substantial portion of patients exhibit resistance to antipsychotics, emphasizing the need for exploring non-pharmacological treatments. In clinical practice, Electroconvulsive therapy (ECT) has been shown to be generally effective in psychosis, but its clinical use sometimes is limited by its cognitive side effects. Magnetic Seizure Therapy (MST) is a novel modification of electroconvulsive therapy (ECT). MST offers the advantages of milder side effects on cognition, a quicker return of orientation, and a shorter duration of post-ictal confusion. A few studies have studied the antipsychotic effect of MST. Therefore, the present study will plan to perform a clinical trial to compare the efficacy of MST treatment plus antipsychotics to antipsychotic medications alone among psychotic disorders in acute phase. In addition, whether MST treatment plus antipsychotics will bring a quicker efficacy response than antipsychotic medications alone is also of important clinical significance. The present trial will plan to administer 10 sessions of MST in 2 weeks, in which the patients will be randomly allocated to either receiving MST+medications or receiving medications alone. After the 2 week's research intervention, all patients will be switched to clinical routine management, but kept under masked clinical assessment for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* (1) meets the diagnostic criteria for schizophrenia or other primary psychotic disorders according to DSM-5;
* (2) age range between 18 and 55 years;
* (3) Positive And Negative Syndrome Scale (PANSS) score≥60;
* (4) to provide informed consent.

Exclusion Criteria:

* (1) have a concomitant severe medical illness;
* (2) are pregnant or intend to get pregnant during the study;
* (3) have a history of DSM-5 diagnosis of substance dependence or abuse within the past three months;
* (4) history of traumatic brain injury (with a screening scale score of 7 or above);
* (5) history of poor response to electroconvulsive therapy or MST;
* (6) have probable dementia based on study investigator assessment; have any significant neurological disorder or condition likely to be associated with increased intracranial pressure or a space occupying brain lesion, e.g., cerebral aneurysm;
* (7) presenting with a medical condition, medication, or laboratory anomaly deemed by the investigator to potentially induce psychotic symptoms, or significant cognitive impairment. (e.g., hypothyroidism with low TSH, rheumatoid arthritis requiring high dose prednisone, or Cushing's disease);
* (8) have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
* (9) a score of 18 or more on the 24-item Hamilton Depression Rating Scale (HAM-D);
* (10) needing ECT treatment immediately due to such dangerous symptoms as suicide, stupor or psychomotor agitation, etc.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Positive and Negative Symptom Scale (PANSS) | Baseline, 1 weeks, 2 weeks, 6 weeks
  measured by Positive and Negative Symptom Scale (PANSS)

SECONDARY OUTCOMES:
Changes in cognition | Baseline, 1 weeks, 2 weeks
  measured by MCCB cognition tests
Changes of ictal EEG feature | during each treatment
  measured by electroencephalogram (EEG)
Changes of cortical inhibition | baseline, 2 weeks
  measured by TMS evoked potentials (TEP)
Changes of brain grey matter | baseline, 2 weeks
  measured by structural MRI images of brain
Changes in 24-item Hamilton Depression Rating Scale (HAM-D) | Baseline, 1 weeks, 2 weeks, 6 weeks
  measured by 24-item Hamilton Depression Rating Scale (HAM-D)
Changes in Hamilton Anxiety Scale (HAMA) | Baseline, 1 weeks, 2 weeks, 6 weeks
  measured by Hamilton Anxiety Scale (HAMA)
Changes in Clinical Global Impression (CGI) scale | Baseline, 2 weeks, 6 weeks
  measured by Clinical Global Impression (CGI) scale
Changes in Global Assessment of Functioning (GAF) scale | Baseline, 2 weeks, 6 weeks
  measured by Global Assessment of Functioning (GAF) scale
Changes in brain gamma band signal | Baseline, 2 weeks
  Gamma band signal will be measured by magnetoencephalogram (MEG)

CONTACTS AND LOCATIONS:
Overall Officials: Jijun Wang, M.D, Ph.D, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang J, Li J, Xu Y, Zhang B, Sheng J, Liu D, Wang W, Yang F, Guo X, Li Q, Zhang T, Tang Y, Jia Y, Daskalakis ZJ, Wang J, Li C. Magnetic Seizure Therapy Compared to Electroconvulsive Therapy for Schizophrenia: A Randomized Controlled Trial. Front Psychiatry. 2021 Nov 25;12:770647. doi: 10.3389/fpsyt.2021.770647. eCollection 2021. PMID 34899429
- [Background] Jiang J, Li Q, Sheng J, Yang F, Cao X, Zhang T, Jia Y, Wang J, Li C. 25 Hz Magnetic Seizure Therapy Is Feasible but Not Optimal for Chinese Patients With Schizophrenia: A Case Series. Front Psychiatry. 2018 May 29;9:224. doi: 10.3389/fpsyt.2018.00224. eCollection 2018. PMID 29896130
- [Background] Daskalakis ZJ, Tamminga C, Throop A, Palmer L, Dimitrova J, Farzan F, Thorpe KE, McClintock SM, Blumberger DM. Confirmatory Efficacy and Safety Trial of Magnetic Seizure Therapy for Depression (CREST-MST): study protocol for a randomized non-inferiority trial of magnetic seizure therapy versus electroconvulsive therapy. Trials. 2021 Nov 8;22(1):786. doi: 10.1186/s13063-021-05730-7. PMID 34749782
- [Background] Daskalakis ZJ, McClintock SM, Hadas I, Kallioniemi E, Zomorrodi R, Throop A, Palmer L, Farzan F, Thorpe KE, Tamminga C, Blumberger DM. Confirmatory Efficacy and Safety Trial of Magnetic Seizure Therapy for Depression (CREST-MST): protocol for identification of novel biomarkers via neurophysiology. Trials. 2021 Dec 11;22(1):906. doi: 10.1186/s13063-021-05873-7. PMID 34895296